CLINICAL TRIAL: NCT06102044
Title: Trial of Zinc Supplements for Young Infants With Clinical Severe Infection in Tanzania
Brief Title: Zinc Supplementation for Young Infants With Clinical Severe Infection in Tanzania
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Christopher Robert Sudfeld, Associate Professor of Global Health and Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB23-0138
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc Supplementation (Experimental): 14-day regimen of twice-daily 5 mg elemental zinc supplements to be taken orally or by enteral feeding tube
  Interventions: Dietary Supplement: Zinc Supplements
- Placebo (Placebo Comparator): 14-day regimen of twice-daily oral placebo supplements to be taken orally or by enteral feeding tube
  Interventions: Dietary Supplement: Placebo Supplements

INTERVENTIONS:
Dietary Supplement: Zinc Supplements — Dispersible zinc citrate tablets
  Arms: Zinc Supplementation
Dietary Supplement: Placebo Supplements — Dispersible placebo tablets
  Arms: Placebo

SUMMARY:
Bacterial infections among young infants, including sepsis, meningitis, and pneumonia, continue to cause a substantial number of deaths globally. Zinc supplementation in combination with standard antibiotic therapy may represent a new intervention to reduce mortality and improve treatment outcomes for young infants with clinical severe infection.

The Investigators will conduct a randomized, double-blind, placebo-controlled trial of zinc supplementation among young infants 0-59 days with severe clinical infection. The trial will enroll 3,250 Tanzanian infants hospitalized with clinical severe infection as defined by WHO Integrated Management of Childhood Illness (IMCI) guidelines. Enrolled infants will receive standard clinical management including antibiotics and will be randomized to receive either a 14-day course of twice-daily 5 mg elemental zinc (10 mg per day) or a matching placebo regimen.

ELIGIBILITY:
Inclusion Criteria:

* Young infants aged 0-59 days
* Diagnosis of clinical severe infection (CSI)
* Ability to feed enterally
* Intend to stay in the study area for 90 days
* Provided informed consent

Exclusion Criteria:

* Prior use of zinc supplements during the current illness
* Receipt of antibiotics for >24 hours before enrollment
* Diarrhea at enrollment
* Signs suggestive of serious illness/condition that is not clinical severe infection
* Previously enrolled in the trial
* Enrolled in other research study

Ages: 0 Days to 59 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3250 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Death | 90 Days
  All-cause infant death
Treatment Failure | From date of randomization until the date of first documented treatment failure or date of death from any cause during the initial hospitalization, whichever comes first, assessed up to 90 days
  A composite endpoint of death during initial period of hospitalization, the need for additional respiratory support (either mechanical ventilation, or positive end expiratory pressure support) or the use of vasoactive medicines to support blood pressure or need to change antibiotics during the initial hospitalization

SECONDARY OUTCOMES:
Death during initial hospitalization | Randomization to the date of initial hospitalization discharge, assessed up to 90 days
  All-cause mortality during initial hospitalization
Duration of initial hospital stay | Randomization to Day 90
  Hours from randomization to initial hospitalization discharge
Duration of signs of clinical severe infection | Randomization to Day 90
  Hours from randomization to the absence of any sign of clinical severe infection
Diarrhea during initial hospital admission | Randomization to the date of initial hospitalization discharge, assessed up to 90 days
  Clinical diagnosis based on three or more loose or watery stools in the past 24 hours
Rate of vomiting related to regimen dosing | Randomization to Day 15
  Vomiting observed by study staff within 30 minutes of regimen dosing
Re-hospitalization | Date of initial hospitalization discharge to Day 90
  Infant admitted and stayed overnight in health facility after being discharged from initial hospitalization
Presence of any sign of possible severe bacterial infection at Day 15 | Day 15
  Presence of a clinical sign of possible severe bacterial infection, including: high body temperature ≥38°C, low body temperature <35.5°C , severe chest indrawing, movement only on stimulation or no movement at all, stopped feeding well or unable to feed at all, or convulsions.
Presence of any sign of possible severe bacterial infection at Day 90 | Day 90
  Presence of a clinical sign of possible severe bacterial infection, including: high body temperature ≥38°C, low body temperature <35.5°C , severe chest indrawing, movement only on stimulation or no movement at all, stopped feeding well or unable to feed at all, or convulsions.
Proportion of Children with Diarrhea at Day 15 or Day 90 | Day 15 and Day 90
  Maternal report of three or more loose or watery stools in the past 24 hours
Infant length-for-age z-score at Day 15 | Day 15
  Infant length-for-age z-score by WHO Child Growth Standards
Infant length-for-age z-score at Day 90 | Day 90
  Infant length-for-age z-score by WHO Child Growth Standards
Infant weight-for-age z-score at Day 15 | Day 15
  Infant weight-for-age z-score by WHO Child Growth Standards
Infant weight-for-age z-score at Day 90 | Day 90
  Infant weight-for-age z-score by WHO Child Growth Standards
Infant weight-for-length z-score at Day 15 | Day 15
  Infant weight-for-length z-score by WHO Child Growth Standards
Infant weight-for-length z-score at Day 90 | Day 90
  Infant weight-for-length z-score by WHO Child Growth Standard
Plasma zinc concentrations at Day 15 | Day 15
  Infant plasma zinc concentration

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Sudfeld, ScD, Principal Investigator — Harvard School of Public Health (HSPH); Christopher P Duggan, MD, Principal Investigator — Harvard School of Public Health (HSPH) and Boston Children's Hospital; Karim P Manji, MD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Manji KP, Somji S, Bakari M, Fawzi WW, Kibwana U, Kisenge R, Kisumuni AS, Liu E, Mafie N, Maleko FA, Salim N, Duggan CP, Sudfeld CR. Efficacy of zinc supplementation for young infants with clinical severe infection in Tanzania: study protocol for a randomised controlled trial. BMJ Paediatr Open. 2025 Aug 14;9(1):e003804. doi: 10.1136/bmjpo-2025-003804. PMID 40813142